CLINICAL TRIAL: NCT00878280
Title: Copy Number Variations, Expression of Inflammatory Cytokines and the Risk of Dementia - A Two-stage Genome-wide Association Study
Brief Title: Copy Number Variations, Inflammatory Cytokines and the Risk of Dementia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yen-Ching Chen, Institute of Preventive Medicine College of Public Health National Taiwan University
Other Study IDs: 200712102R-1
Record Dates: First submitted 2008-08-31; First posted 2009-04-08 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 1:control(healthy subjects)
- 2: 2:case(dementia patients)

SUMMARY:
Assess the association of copy number variation (CNV) and inflammatory cytokine with the risk of dementia.

DETAILED DESCRIPTION:
This is a hospital-based case-control study. We plan to assess the association of CNV and inflammatory cytokine with the risk of dementia. Hopefully to find some genetic biomarkers to identify the risk of dementia at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* hospital recruited dementia patients and controls

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: hospital recruited dementia patients and controls
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-08; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Dementia | Aug 2008-July 2011

CONTACTS AND LOCATIONS:
Overall Officials: yen-ching chen, ScD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan